CLINICAL TRIAL: NCT06445400
Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of BL-M07D1, BL-M07D1+Pertuzumab and BL-M07D1+Pertuzumab+Docetaxel as First-line Treatment in Patients With Unresectable Locally Advanced or Metastatic HER2-positive Breast Cancer
Brief Title: A Study of BL-M07D1, BL-M07D1+Pertuzumab and BL-M07D1+Pertuzumab+Docetaxel in Patients With Unresectable Locally Advanced or Metastatic HER2-positive Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M07D1-205
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — pertuzumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants received BL-M07D1, BL-M07D1+Pertuzumab and BL-M07D1+ Pertuzumab+Docetaxel in the first cycle (3 weeks). Participants who had a clinical benefit could receive additional cycles of additional treatment. Administration will be discontinued because of disease progression or intolerable toxicity or for other reasons.
  Interventions: Drug: BL-M07D1; Drug: Pertuzumab; Drug: Docetaxel

INTERVENTIONS:
Drug: BL-M07D1 — Administration by intravenous infusion for a cycle of 3 weeks.
Drug: Pertuzumab — Administration by intravenous infusion for a cycle of 3 weeks.
Drug: Docetaxel — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This study is a phase II clinical trial to evaluate the safety and efficacy of BL-M07D1, BL-M07D1+Pertuzumab and BL-M07D1+Pertuzumab+Docetaxel as first-line treatment in patients with unresectable locally advanced or metastatic HER2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Gender is not limited;
3. Age ≥18 years old and ≤75 years old;
4. Expected survival time for 3 months or more;
5. Patients with histologically and/or cytologically confirmed unresectable locally advanced or metastatic HER2-positive breast cancer;
6. Consent to provide archived tumor tissue samples or fresh tissue samples from the primary or metastatic lesions;
7. At least one measurable lesion meeting the RECIST v1.1 definition was required;
8. Physical condition score ECOG 0 or 1 ;
9. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. No blood transfusion, no colony-stimulating factor, and no albumin are allowed within 14 days before the first use of the study drug, and the organ function level must meet the requirements;
12. Blood coagulation function: international standardization ratio (INR) 1.5 or less, and the part activated clotting time (APTT) live enzymes acuities were 1.5 x ULN;
13. Urinary protein ≤2+ or ≤1000mg/24h;
14. Fertile female subjects, or male subjects with fertile partners, must use highly effective contraception from 7 days before the first dose until 7 months after the end of the dose. Female subjects of childbearing potential had to have a negative serum pregnancy test within 7 days before the first dose.

Exclusion Criteria:

1. Received chemotherapy with mitomycin C and nitrosourea within 6 weeks before the first dose, received surgery within 4 weeks before the first dose, and received endocrine therapy within 2 weeks before the first dose;
2. Patients with locally advanced or metastatic disease who have received previous systemic therapy;
3. Had received prior ADC drug therapy with camptothecin derivative as toxin;
4. Screening within the first half of the serious heart, cerebrovascular disease;
5. Complicated with pulmonary diseases leading to severe impairment of lung function;
6. A history of ILD/interstitial pneumonia requiring steroid therapy, current ILD/interstitial pneumonia, or suspected ILD;
7. QT prolongation, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
8. Other primary malignancies diagnosed within 5 years before the first dose;
9. Poorly controlled hypertension;
10. Patients with active central nervous system metastases;
11. Need treatment intervention of unstable thrombotic events, except infusion related thrombosis;
12. Patients with a history of allergy to recombinant humanized antibodies or to any excipients of the trial drug;
13. Had received more than the following cumulative doses of anthracyclines;
14. Systemic corticosteroids or immunosuppressive agents were required within 2 weeks before study dosing;
15. Patients with massive or symptomatic effusions or poorly controlled effusions;
16. Severe systemic infection within 4 weeks before screening;
17. Active autoimmune and inflammatory diseases;
18. Human immunodeficiency virus antibody positive, active hepatitis B virus infection or hepatitis C virus infection;
19. Previous history of allogeneic stem cell, bone marrow or organ transplantation;
20. A history of severe neurological or psychiatric illness;
21. Pregnancy or lactation women;
22. Patients who were deemed by the investigator to be ineligible for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-M07D1.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-M07D1 to the first date of either disease progression or death, whichever occurs first.
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M07D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M07D1.

CONTACTS AND LOCATIONS:
Overall Officials: Herui Yao, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Qiang Liu, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China